CLINICAL TRIAL: NCT02039635
Title: A Study of Korean Red Ginseng for Evaluation of Improvement of Cancer-related Fatigue in Patients With Colorectal Cancer With Chemotherapy: A Randomized, Double-blind, Placebo-Controlled, Parallel, Multicenter Trial
Brief Title: Korean Red Ginseng in Treating Patients With Fatigue Caused by Chemotherapy for Colorectal Cancer
Acronym: KRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Ginseng Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KGC-S-02
Record Dates: First submitted 2013-12-16; First posted 2014-01-17 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: cancer; cancer related fatigue; Korean red ginseng; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Korean Red Ginseng (Experimental): Patients receive oral Korean Red Ginseng twice daily for 16 weeks. Treatment repeats every 4 weeks for 4 courses.
  Intervention: Dietary Supplement: Korean Red Ginseng
  Interventions: Dietary Supplement: Korean Red Ginseng
- Placebo (Placebo Comparator): Patients receive oral placebo twice daily for 16 weeks. Treatment repeats every 4 weeks for 4 courses.
  Intervention: Other: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — Given Orally
  Arms: Korean Red Ginseng
Dietary Supplement: Placebo — Given Orally
  Arms: Placebo

SUMMARY:
Korean Red Ginseng may improve fatigue in healthy subject. It is not yet known whether Korean Red Ginseng is effective compared with a placebo in chemotherapy.

The purpose of this study is to determine whether Korean Red Ginseng is effective in the treatment of the fatigue from colorectal cancer with chemotherapy.(modified FOLFOX-6)

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* Person who agreed to participate in this study and signed voluntarily on the written informed consent form
* Person who is confirmed as colorectal cancer through histological and image diagnosis and scheduled for adjuvant or palliative therapy with mFOLFOX-6 regimen
* Fertile patients with negative pregnancy test confirmed and who has agreed to use effective contraception
* Person who is able to fully communicate with the physician about his/her fatigue status and is able to completely fill out the questionnaires
* Life expectancy more than 6 months
* Performance status of ECOG grade 0~1
* Hb ≥ 9g/dL
* Person with moderate liver function (AST, ALT ≤ 2.5 × ULN)
* Person with moderate renal function (Cr ≤ 1.5 × ULN)

Exclusion Criteria:

* Pregnant or nursing women
* Primary brain cancer, brain metastases or other CNS malignancy, including CNS lymphoma
* No controlled pain despite the use if analgesics.
* Person showing hypothyroidism despite the hormone treatment
* Person with insomnia despite an appropriate treatment
* No controlled hypertension (DBP >100mmHg or SBP >160mmHg)
* Person who has experience of hypersensitivity to the trial drug (ginseng) components
* Person with autoimmune disorders (Multiple sclerosis, Lupus, rheumarthritis etc.)
* Person who is alcoholic dependent or has psychiatric disorder
* Person who has cognitive or psychiatric problems
* Person who has an experience of chemotherapy agents use 6 months before a screening visit
* Person who had a surgery 2 weeks before a screening visit
* Person who had taken herbal medicinal product (including Chinese medicine) 4 weeks before the screening visit
* Person who has medical status that is judged to affect the result or who is judged as inappropriate for the study by the physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of Brief Fatigue Index (BFI) on the intake trial drugs up to 16 weeks | From Baseline up to 16 weeks

SECONDARY OUTCOMES:
Area Under Curve (AUC) of Brief Fatigue Index (BFI) on the intake of trial drugs up to 8 weeks | From Baseline up to 8 weeks
Change in Functional Assessment of Chronic Illness Therapy-Fatigue Trial Outcome Index (FACIT-F TOI) after 8 and 16 weeks of trial drug intake | Baseline, 8 and 16 weeks
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) total score after 8 and 16 weeks of trial drug in take | Baseline, 8 and 16 weeks
The percentage of subjects whom the Functional Assessment of Cancer Therapy-General (FACT-G) score decreased more than 20 scores after 8 and 16 weeks of trial drug intake | Baseline, 8 and 16 weeks
Change in blood cytokine (IL-1, IL-6, TNF-alpha) level after 16 weeks of trial drug intake | Baseline, 16 weeks
Change in blood cortisol level after 16 weeks of trial drug intake | Baseline, 16 weeks
Perceived Stress Scale (PSS) change after 16 weeks of trial drug intake | Baseline, 16 weeks
adverse events | Baseline, 8 and 16 weeks
  * Voluntary reports of adverse events and collected reports of adverse events (agitation, anxiety, headache, insomnia, vomiting)
  * Laboratory and physical test
  * ECOG performance
  * ECG

OTHER OUTCOMES:
Tumor response after 8 and 16 weeks of trial drug intake | Baseline, 8 and 16 weeks
Progressive-free survival (PFS) | up to 16 weeks
Change in blood cytokine(IL-2, IL-8, IL-10) level after 16 weeks of trial drug intake | Baseline, 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Ginseng Corporation, Shinseongdong, Daejeon, South Korea